CLINICAL TRIAL: NCT03329781
Title: Modulation of Endotoxaemia Via Curcumin Intake in Healthy Overweight Adults
Brief Title: ENDOCUR - Modulation of Endotoxaemia Via Curcumin Intake in Healthy Overweight Adults
Acronym: ENDOCUR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Emilie Combet, Senior Lecturer, University of Glasgow
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 200130089
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Overweight
Keywords: Endotoxaemia, Curcumin.
MeSH Terms: conditions — Overweight; Endotoxemia

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Trial (Experimental): 350 mg of BCM-95, 1 capsule per day, for 21 days.
  Interventions: Dietary Supplement: BCM-95
- Control (Placebo Comparator): 350 mg of starch, 1 capsule per day, for 21 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: BCM-95 — Consuming 1 capsule of BCM-95 per day.
  Other Names: Bio-Curcumin
  Arms: Trial
Dietary Supplement: Placebo — Consuming 1 placebo capsule per day
  Arms: Control

SUMMARY:
Chronic diseases such as diabetes, cardiovascular diseases and cancer are a major burden on the Scottish population. Obesity and inflammation have strong links to these diseases. One of the mechanisms explaining the relationship between low-grade inflammation and excess weight is "endotoxaemia". We wish to study this phenomenon, when small components coming from our gut bacteria can pass into the bloodstream, raising the body's defences. Diet can modulate endotoxaemia. In this study, we propose to use curcumin, in a capsule form, to modulate endotoxaemia. Curcumin comes from turmeric, which is widely used as a spice. In this study, we want to test the effect of consuming curcumin extract to the composition of the gut microbiota, post-meal endotoxaemia, and inflammatory markers in blood.

ELIGIBILITY:
Inclusion Criteria:

- BMI > 25 kg/m2.

Exclusion Criteria:

* having chronic inflammatory or autoimmune disease, gastrointestinal complaints or known biliary obstruction (past and present)
* use of anti-inflammatory drugs 2 weeks before the start of the study
* use of antibiotics during the 12 weeks preceding the trial
* pregnancy
* lactation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Level of endotoxin in plasma. | 21 days